CLINICAL TRIAL: NCT05598619
Title: Effect of Colon Delivered Vitamin C on Gut Microbiota and Related Health Biomarkers in Healthy Older Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: DSM Nutritional Products, Inc. (Industry)
Collaborators: Atlantia Food Clinical Trials (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: 020-11-11-VITC
Record Dates: First submitted 2022-10-25; First posted 2022-10-28 (Actual); Last update posted 2024-08-22 (Actual); Status verified 2024-08

CONDITIONS: Quality of Life
Keywords: microbiota; vitamin; short chain fatty acids
MeSH Terms: interventions — Ascorbic Acid; microcrystalline cellulose

STUDY DESIGN:
Intervention Model Description: Randomized, double-blind, placebo-controlled, parallel trial
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Low dose (Experimental): Daily dose of 80 mg Vitamin C (Ascorbic acid) once a day for 12 weeks
  Interventions: Dietary Supplement: Vitamin C
- Mid dose (Experimental): Daily dose of 200 mg Vitamin C (Ascorbic acid) once a day for 12 weeks
  Interventions: Dietary Supplement: Vitamin C
- High dose (Experimental): Daily dose of 500 mg Vitamin C (Ascorbic acid) once a day for 12 weeks
  Interventions: Dietary Supplement: Vitamin C
- Placebo (Placebo Comparator): One capsule of 570 mg (consisting microcrystalline cellulose) once a day for 12 weeks
  Interventions: Other: placebo

INTERVENTIONS:
Dietary Supplement: Vitamin C — Colon delivered vitamin C (ascorbic acid) for 12 weeks
  Other Names: Ascorbic acid
  Arms: High dose; Low dose; Mid dose
Other: placebo — Colon delivered placebo once a day for 12 weeks
  Other Names: Microcrystalline cellulose
  Arms: Placebo

SUMMARY:
Recent studies have shown that many vitamins, if consumed in high daily dosages or delivered to the colon, can modulate the gut microbiota and their metabolites. In parallel, gut microbiota imbalances are linked to diseases, e.g., obesity, type 2 diabetes, cardiovascular disease, autoimmune diseases, and intestinal inflammatory diseases. Therefore, vitamin administration could offer health benefits beyond those traditionally considered for these nutrients. Earlier, our group investigated the effect of colon-delivered vitamins A, B2, C, D, and E on the gut microbiota using a human clinical trial and showed that vitamin C, B2, and D modulates the human gut microbiome in terms of metabolic activity and bacterial composition. The most distinct effect was that of vitamin C, which significantly increased microbial alpha diversity and fecal short-chain fatty acids compared to the placebo. However, the dose-dependent and combined effect of colon-delivered vitamins on the microbial community and its subsequent impact on host health is unknown. This study will investigate the effect of colon-delivered vitamin C (three dosages) on the gut microbiome.

ELIGIBILITY:
Inclusion Criteria:

1. Participants must be willing and able to give written informed consent and to understand, to participate, and to comply with the clinical study requirements.
2. Between 50 and 70 years of age.
3. Has a BMI of between 18.5 - 30 Kg/m2.
4. Participants have had a stable body weight (≤5 % change) over the past 3-months.
5. Is in general good health, as determined by interview and vital signs (blood pressure, heart rate, pulse) by the investigator.
6. Willing to avoid consuming gut microbiome modulating dietary supplements, prebiotic, probiotic, or fibre-rich supplements, and, within 4 weeks prior to the baseline visit, until the end of the study.
7. Maintain current level of physical activity.
8. Willing to consume the investigational product daily for the duration of the study.
9. Female participants in menopause for at least the last one year.

Exclusion Criteria:

1. Are hypersensitive to any of the components of the test product.
2. Has taken antibiotics within the previous 3 months prior to Baseline (Visit 2).
3. Is currently using systemic steroids, systemic antibiotics, proton pump inhibitors, H2 blocker, antacid, metformin, or immunosuppressant medication.
4. Participant has a history of drug and/or alcohol abuse at the time of enrolment (Drinks more than nationally recommended units per week (>11 units for women; >17 units for men); Is currently in treatment for alcohol/substance abuse; Has been diagnosed with alcohol/substance abuse disorder).
5. Is a smoker or vaper.
6. Vegetarian or vegan.
7. Has made any major dietary changes in the past 3 months prior to Baseline (Visit 2).
8. Planned major changes in the lifestyle (i.e., diet, dieting, exercise level, significant travel) during the duration of the study.
9. Has a currently active eating disorder.
10. Has food allergies or other issues with foods that would preclude the intake of the study products, as determined by the study investigator.
11. Is having a typical fibre intake >30 g fibre/day.
12. Has an active gastrointestinal disorder or previous gastrointestinal surgery, which in the opinion of the investigator would impact the study outcomes.
13. If taking chronic medications (e.g., anti-hypertensive medications), they must have been taking the product for at least two months to screening and agree to maintain the same dosage throughout the study.
14. Has severe or uncontrolled type 2 diabetes, psychiatric disorder, gastrointestinal disease (i.e., diarrhoea, Crohn's disease, ulcerative colitis, IBS, diverticulosis, stomach or duodenal ulcers respiratory or cardiac illness or any other condition which in the opinion of the investigator would impact the study outcomes.
15. Has a current or history of any gastrointestinal cancer
16. Are severely immunocompromised (HIV positive, transplant patient, on anti-rejection medications, on a steroid for >30 days, or chemotherapy or radiotherapy with the last year).
17. Experiences alarm features such as weight loss, rectal bleeding, a recent change in bowel habit (<3 months).
18. Have a current malignant disease or any concomitant end-stage organ disease.
19. Individuals who, in the opinion of the investigator are considered to be poor attendees or unlikely for any reason to be able to comply with the trial.
20. Participants may not be receiving treatment involving experimental drugs. If the participant has been in a recent experimental trial, these must have been completed not less than 60 days prior to this study.
21. Participants who have undergone intensive skin treatments (e.g. laser treatment or skin related surgery) in the last 3 months.
22. If taking any dietary supplements or medications known to affect skin health or other trial measures (resveratrol, ginkgo biloba, ginseng, fruit powder extracts and DHA).
23. Has a skin condition likely to interfere with skin assessments (e.g., eczema, dermatitis, any open skin wounds, reactive and sensitive skin).

    -

Ages: 50 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 264 (Actual)
Dates: Start 2022-07-01 (Actual); Primary Completion 2023-03-13 (Actual); Study Completion 2023-03-13 (Actual)

PRIMARY OUTCOMES:
Microbial metabolites measured as short-chain fatty acid content in faeces, at baseline and at week 12. | from baseline to 12 weeks
  To assess the changes of microbial metabolites from baseline to 12 weeks supplementation of three different doses of colon delivered vitamin C to compare the changes to placebo.

SECONDARY OUTCOMES:
Faecal microbial composition and diversity | from baseline to 12 weeks
  Faecal microbial composition at phylum, genus, and species levels, and alpha and beta diversity indices at the genus and species level as measured by metagenomic based profiles at baseline and at week 12.
Intestinal inflammation | from baseline to 12 weeks
  Intestinal inflammation as assessed by faecal calprotectin at baseline and at week 12.
Intestinal barrier integrity | from baseline to 12 weeks
  Intestinal barrier integrity as assessed by sCD14 at baseline and at week 12.
Oxidative stress in blood | from baseline to 12 weeks
  Oxidative stress level measured as free thiol content in blood at baseline and at week 12.
Inflammatory status in blood | from baseline to 12 weeks
  Systemic inflammation measured as high sensitive C reactive protein (hs-CRP) in blood at baseline and at week 12.
Gastrointestinal symptoms and quality of life | from baseline to 12 weeks
  Gastrointestinal symptoms and quality of life as assessed by Gastrointestinal Symptom Rating Scale (GSRS) and short form survey-36 (SF-36) questionnaires at baseline and at week 12.
Stool consistency | from baseline to 12 weeks
  Stool consistency (Bristol Stool Scale), as reported in the daily eDiary app (at baseline and week 12).
Stool frequency | from baseline to 12 weeks
  Stool frequency, as reported in the daily eDiary app (at baseline and week 12).
Systemic vitamin status | from baseline to 12 weeks
  The concentration of vitamin C in blood at baseline and at week 12.
Faecal pH | from baseline to 12 weeks
  Faecal pH at baseline and at week 12.
Faecal microbial composition and diversity | from baseline to 4 weeks
  Faecal microbial composition at phylum, genus, and species levels, and alpha and beta diversity indices at the genus and species level as measured by metagenomic based profiles at baseline and at week 4.
Microbial metabolites | from baseline to 4 weeks
  Faecal microbial metabolites measured as short-chain fatty acid content at baseline and week 4.

CONTACTS AND LOCATIONS:
Overall Officials: Prof Timothy Dinan, Principal Investigator — Cork University Hospital
Locations (1):
- Atlantia Food Clinical Trials, 1st Floor, Block C, Heron House, Blackpool Retail Park, Cork, Cork, Ireland